CLINICAL TRIAL: NCT03149679
Title: Treatment of Patients With Metastatic Colorectal Cancer Harboring TP53 Mutations With Dose-dense Cyclophosphamide - the p53 Colorectal Cancer Trial
Brief Title: The p53 Colorectal Cancer Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was discontinued after the first pre-planned interim analysis due to insufficient response rates.
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/1637
Record Dates: First submitted 2017-03-14; First posted 2017-05-11 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer Metastatic; Colorectal Cancer Stage IV; TP53 Gene Mutation
Keywords: Cyclophosphamide; Colorectal Cancer Metastatic; TP53 Gene Mutation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Single center, open labeled, phase 2 clinical trial, where patients are selected for treatment based on upfront TP53 mutation status; i.e. only patients with TP53 mutated tumors may be included in the single treatment arm. The informed consent, however needs to be signed prior to a biopsy for TP53 mutation analyses; thus, all patients are formally enrolled in the study prior to tissue collection, and the full population tested will be accounted for despite the fact that only patients with TP53 mutated tumors may enter the single treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cyclophosphamide arm (Experimental): Dose dense cyclophosphamide (1800 Mg/m2) administered intravenously every second week.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — Chemotherapy
  Other Names: Sendoxan

SUMMARY:
Single center, open labeled, phase 2 clinical trial, where patients with metastatic colorectal cancer are selected for treatment with dose dense Cyclophosphamide every second week based on TP53 mutation status; i.e. only patients with TP53 mutated tumors may be included in the treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer patients for whom conventional therapy has failed; defined as 2 lines of chemotherapy including oxaliplatin or irinotecan- containing regimens as well as an EGFR inhibitor if applicable.
* Tumor lesion suitable for biopsy
* Age >18 years
* Clinically or radiologically measurable tumor deposits according to the RECIST criteria
* WHO performance status 0-1
* Radiology studies (CT thorax/abdomen/pelvis) and echo cor and ECG must be performed within 28 days prior to registration.
* Before patient registration in the trial, written informed consent must be given according to national and local regulations.
* Blood test requirements:

Neutrophils > 1.0 e9/L Platelets > 75 e9/L Bilirubin < 20 µmol / L. Serum creatinine < 1.5 x ULN

Exclusion Criteria:

* Co-morbidity including, but not limited to, impaired renal-, liver or bone marrow function, that based on the assessment of the treating physician, may preclude the use of cyclophosphamide at actual doses.
* Known hypersensitivity to the study drug, its metabolites or any excipients in the infusion solution.
* Psychological, familial, sociological or geographical condition(s) potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Pregnant or lactating patients cannot be included.
* Clinical evidence of serious coagulopathy. Prior arterial/venous thrombosis or embolism does not exclude patients from inclusion, unless patient is considered unfit by study oncologist.
* Patient not able to give an informed consent or comply with study regulations as deemed by study investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 4 months
  Partial response (PR) or complete response (CR) as defined by the RECIST criteria

SECONDARY OUTCOMES:
Possible molecular markers of therapy response/resistance and survival outcome beyond TP53 mutations will be examined. | 10 years
  Tissue and blood sampling at baseline and whenever treatment is changed
Number of patients with treatment response among patients harboring TP53 mutations belonging to particular mutation subgroups | 10 years
  Tissue and blood sampling at baseline and whenever treatment is changed
Clinical benefit rate (CBR) | 5 years
  Stable disease (SD) >6 months, PR or CR
Recurrence-free and overall survival, compared to historical data | All patients will be followed for 5 years or until death to record survival outcome
  Survival analyses
Safety and tolerability of the study treatment including recording of number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Every second week during the treatment period from start of treatment, and thereafter every second month for 5 years or until death
  Clinical examination and blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Inger Marie Løes, MD PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No